CLINICAL TRIAL: NCT01075880
Title: Post-Authorization Observational Study to Evaluate Cognition and Fatigue in RRMS Patients Treated With Rebif
Brief Title: Post-Authorization Observational Study to Evaluate Cognition and Fatigue in Relapsing-remitting Multiple Sclerosis (RRMS) Patients Treated With Rebif®
Acronym: SKORE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck spol.s.r.o., Czech Republic (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-519
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Rebif; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rebif (Interferon beta-1a) — The treatment to be administered is interferon beta-1a on prescription, used as per SmPC, i.e. both doses 22 and 44 mcg s.c. tiw, and the titration pack 8.8 mcg and 22 mcg s.c. tiw when initiating the therapy.
  Other Names: Rebif

SUMMARY:
The study is planned to evaluate the cognitive functions in subjects with RRMS treated with interferon beta-1a, and its relationship to the fatigue and neurological dysfunction status.

DETAILED DESCRIPTION:
Besides the motor and sensory dysfunctions, the progression of cognitive decline is a frequent manifestation of RRMS. Fatigue is another important symptom of MS, and can negatively affect subject's Quality of life (QoL) and socio-economic functioning, including the ability to work, independent of the direct effects of disability. This is a phase IV observational, non-interventional, prospective, multicentric study to evaluate cognition in RRMS subjects treated with Rebif and its relationship to the fatigue and neurological dysfunction status. The study plans to enroll 300 subjects, across 14 centres in Czech Republic, who will be prescribed with Rebif according to its summary of product characteristics (SmPC). Assessment of cognitive and fatigue status will be done at baseline and follow-up visits at Months 3, 6, 12, 24. Subjects will be selected using the convenience method following the non-probability sampling.

OBJECTIVES

Primary Objective:

* To assess changes of cognition [measured by Paced Auditory Serial Addition Test (PASAT)] in RRMS subjects treated with Rebif

Secondary Objectives:

* To assess changes of fatigue [measured by Fatigue Descriptive Scale (FDS)] in RRMS subjects treated with Rebif
* To assess a correlation between cognition, fatigue and neurological status in RRMS subjects treated with Rebif
* To assess a relationship between Rebif dosage [22 mcg vs 44 mcg thrice a week (tiw)] and cognition (PASAT)
* To assess a relationship between Rebif dosage (22 mcg vs 44 mcg tiw) and fatigue (FDS)
* To assess adherence to Rebif treatment
* To explore the use of antidepressive and antifatigue medicaments

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with RRMS
* Subjects eligible for treatment with Rebif as per SmPC, the Czech local guidelines and the actual Health insurance policy.
* Subjects 18-65 years of age
* Subjects with EDSS score < 4
* Subjects who are willing and able to give informed consent

Exclusion Criteria:

* Treatment with Rebif for more than 24 months prior the informed consent form has been obtained.
* Subjects with history of hypersensitivity to natural or recombinant interferon-β, or to any excipients
* Female subject who is pregnant or breast feeding and/or planning to become pregnant
* Subjects with current severe depression and/or suicidal ideation
* Any contraindication for Rebif therapy as per SmPC
* Subjects with severe disability and/or any neurologic or psychiatric condition that may interfere with test performance
* Prior treatment with interferon beta-1a i.m. or interferon beta-1b or glatiramer acetate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with RRMS prescribed with Rebif across 14 centres in Czech Republic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with decreased/increased/stable cognition status (PASAT) | Baseline vs Month 6 - 12 - 24

SECONDARY OUTCOMES:
Percentage of subjects with decreased/increased/stable fatigue (FDS) | Baseline vs Month 6- 12 - 24
Relationship between the cognition status, the fatigue status and the EDSS status | Baseline, Month 6- 12 - 24
Relationship between the Rebif dosage used with cognition and fatigue status | Baseline, Month 6- 12 - 24
Proportion of relapse-free subjects | Month 3 - 6 - 12 - 24
Proportion of subjects with defined EDSS changes (decrease; no change; increase of 0.5 - 1.0; 1.5 - 2.0; 2.5 - 3.0; 3.0 or more points, respectively) | Month 6 - 12 - 24
Proportion of subjects without either relapse, EDSS progression, cognition status decrease and fatigue increase | Month 6 - 12- 24
Number of Rebif doses not taken since the last study visit, and the reason of dose not taken | Month 3 - 6 - 12 - 24
Proportion of subjects using the antidepressive or antifatigue medication | Baseline, Month 3 - 6 - 12 - 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck spol.s.r.o., Czech Republic
Locations (13):
- Czechia (13):
  - Neurologicka klinika FNBB, Brno
  - Neurologicka klinika, Fakultní nemocnice U Sv. Anny, Brno
  - Neurologicke oddeleni KN., České Budějovice
  - Neurologicka klinika Fakultní nemocnice, Hradec Králové
  - Neurologicka klinika Fakultní nemocnice, Motol
  - Neurologicka klinika, Fakultní nemocnice, Olomouc
  - Neurologicka klinika Fakultní nemocnice, Ostrava
  - Neurologicke oddeleni KN, Pardubice
  - Neurologicka klinika Fakultní nemocnice, Pilsen
  - Neurologicka klinika FNKV, Prague
  - Neurologicka klinika, Fakultní Thomayerovy nemocnice, Prague
  - Neurologicke oddeleni NsP, Teplice
  - Neurologicke oddeleni, Baťova nemocnice, Zlín